CLINICAL TRIAL: NCT02470364
Title: Translation, Cross-cultural Adaptation and Validation of the MGQOL-15-F
Acronym: MGQOL-15-F
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: MGQOL-15
Record Dates: First submitted 2015-06-10; First posted 2015-06-12 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2014-10

CONDITIONS: Myasthenia Gravis
Keywords: Myasthenia gravis; Quality of life
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to translate and culturally adapt the MGQOL-15 (health-related quality of life scale for myasthenia gravis) for use with French-speaking patients in France and to evaluate its psychometric properties to ensure reliability and validity.

DETAILED DESCRIPTION:
It is a translation and validation of a quality of life scale.

Step 1: Translation and cultural adaptation (Forward and back translation, committee review, pre-testing with 10 patients for content and face validity).

Step 2 : Psychometric testing : Test-retest with a 2 day interval, correlation with clinical scores - the Myasthenic Muscle Score and the (MG-ADL) score and with a global quality of life score (WHOQOL-BREF).

ELIGIBILITY:
Inclusion Criteria:

* Auto-immune myasthenia gravis
* Age ≥ 18 years old
* Clinical Classification (MGFA) I-IV
* French speaking

Exclusion Criteria:

* cognitive or visual impairment which would limit the capacity to fill out the MGQOL-15-F

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with auto-immune myasthenia gravis
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Perceived quality of life measured via the MGQOL-15-F (French version of the MGQOL-15), a myasthenia-specific quality of life auto-questionnaire | 3 days

SECONDARY OUTCOMES:
Global quality of life evaluated via the WHOQOL-BREF scale | 1 day
Clinical evaluation : Myasthenic Muscle Score | 1 day
Disease severity assessed via the Myasthenic Muscle Score | 1 day
Impact of symptoms on daily activities and daily life using the MG-ADL score | 1day

CONTACTS AND LOCATIONS:
Overall Officials: Simone Birnbaum, Physiotherapist, Principal Investigator — Institute of Myology, La Pitié-Salpêtrière Hospital, 75013 Paris, France
Locations (1):
- Institute of Myology, La Pitié-Salpêtrière Hospital, Paris, France